CLINICAL TRIAL: NCT04234919
Title: A Longitudinal Study of Donor-Derived Cell Free DNA in Lung Transplant
Brief Title: Longitudinal Study of Cell Free DNA in Lung Transplant
Acronym: LoSt
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: 19-2946
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Lung Transplant Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consented adult lung transplant recipients

SUMMARY:
Lung transplant is a viable treatment strategy for many with end-stage lung diseases. Despite advances in both the surgical and medical management, lung transplant recipients experience episodes of allograft insult and injury that lead to dysfunction and ultimately contribute to graft failure. The primary noninvasive tool for monitoring the lung allograft, pulmonary function testing, is neither sensitive nor specific for lung allograft injury which makes the management of lung transplant recipients particularly challenging. A decline in pulmonary function tests prompts invasive procedures such as bronchoscopy with transbronchial lung biopsy to diagnose the cause of allograft injury, although this, too, is not 100% sensitive, and oftentimes patients are treated empirically for rejection when no other etiology for lung function decline is identified. Empiric treatment prompted by extrapulmonary drivers of decline in lung function may result in inappropriate exposure to risks of augmented immunosuppression. The purpose of this study is to determine to what extent monitoring of donor-derived cell free DNA in lung transplant recipients can be used as a marker of lung injury and stability.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Actively listed or have recently had a double lung transplant
* Participant is willing and able to provide informed consent

Exclusion Criteria:

* Prior organ transplantation
* Transplantation performed in the setting of hospitalization for acute illness or decompensation
* Unable or unwilling to consent for enrolment
* Single lung transplant recipient
* Consideration for multi-organ transplantation
* Pregnant women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with end stage lung disease who are placed on the lung transplant waitlist for consideration of a bilateral transplant at the University of Colorado lung transplant program will be recruited for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Relationship | 12 Months
  Determine the relationship between donor derived cell free DNA and lung allograft function during the first year after lung transplant.

SECONDARY OUTCOMES:
Quantitative Assessments | 12 Months
  Quantitative assessments of dd-cfDNA obtained at pre-specified timepoints post-transplant compared to clinical events (PGD scores, detection of allograft dysfunction, rejection, or infection).

CONTACTS AND LOCATIONS:
Overall Officials: Alice L Gray, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chambers DC, Cherikh WS, Goldfarb SB, Hayes D Jr, Kucheryavaya AY, Toll AE, Khush KK, Levvey BJ, Meiser B, Rossano JW, Stehlik J; International Society for Heart and Lung Transplantation. The International Thoracic Organ Transplant Registry of the International Society for Heart and Lung Transplantation: Thirty-fifth adult lung and heart-lung transplant report-2018; Focus theme: Multiorgan Transplantation. J Heart Lung Transplant. 2018 Oct;37(10):1169-1183. doi: 10.1016/j.healun.2018.07.020. Epub 2018 Aug 11. No abstract available. PMID 30293613
- [Background] Glanville AR, Aboyoun CL, Havryk A, Plit M, Rainer S, Malouf MA. Severity of lymphocytic bronchiolitis predicts long-term outcome after lung transplantation. Am J Respir Crit Care Med. 2008 May 1;177(9):1033-40. doi: 10.1164/rccm.200706-951OC. Epub 2008 Feb 8. PMID 18263803
- [Background] Hopkins PM, Aboyoun CL, Chhajed PN, Malouf MA, Plit ML, Rainer SP, Glanville AR. Association of minimal rejection in lung transplant recipients with obliterative bronchiolitis. Am J Respir Crit Care Med. 2004 Nov 1;170(9):1022-6. doi: 10.1164/rccm.200302-165OC. Epub 2004 Aug 5. PMID 15297270
- [Background] Khalifah AP, Hachem RR, Chakinala MM, Yusen RD, Aloush A, Patterson GA, Mohanakumar T, Trulock EP, Walter MJ. Minimal acute rejection after lung transplantation: a risk for bronchiolitis obliterans syndrome. Am J Transplant. 2005 Aug;5(8):2022-30. doi: 10.1111/j.1600-6143.2005.00953.x. PMID 15996255
- [Background] Morrell MR, Pilewski JM, Gries CJ, Pipeling MR, Crespo MM, Ensor CR, Yousem SA, D'Cunha J, Shigemura N, Bermudez CA, McDyer JF, Zeevi A. De novo donor-specific HLA antibodies are associated with early and high-grade bronchiolitis obliterans syndrome and death after lung transplantation. J Heart Lung Transplant. 2014 Dec;33(12):1288-94. doi: 10.1016/j.healun.2014.07.018. Epub 2014 Aug 23. PMID 25443870
- [Background] Kulkarni HS, Bemiss BC, Hachem RR. Antibody-mediated Rejection in Lung Transplantation. Curr Transplant Rep. 2015 Dec;2(4):316-323. doi: 10.1007/s40472-015-0074-5. Epub 2015 Sep 30. PMID 27896040
- [Background] Verleden GM, Glanville AR, Lease ED, Fisher AJ, Calabrese F, Corris PA, Ensor CR, Gottlieb J, Hachem RR, Lama V, Martinu T, Neil DAH, Singer LG, Snell G, Vos R. Chronic lung allograft dysfunction: Definition, diagnostic criteria, and approaches to treatment-A consensus report from the Pulmonary Council of the ISHLT. J Heart Lung Transplant. 2019 May;38(5):493-503. doi: 10.1016/j.healun.2019.03.009. Epub 2019 Apr 3. No abstract available. PMID 30962148
- [Background] Glanville AR, Verleden GM, Todd JL, Benden C, Calabrese F, Gottlieb J, Hachem RR, Levine D, Meloni F, Palmer SM, Roman A, Sato M, Singer LG, Tokman S, Verleden SE, von der Thusen J, Vos R, Snell G. Chronic lung allograft dysfunction: Definition and update of restrictive allograft syndrome-A consensus report from the Pulmonary Council of the ISHLT. J Heart Lung Transplant. 2019 May;38(5):483-492. doi: 10.1016/j.healun.2019.03.008. Epub 2019 Apr 3. No abstract available. PMID 31027539
- [Background] Glanville AR. Bronchoscopic monitoring after lung transplantation. Semin Respir Crit Care Med. 2010 Apr;31(2):208-21. doi: 10.1055/s-0030-1249117. Epub 2010 Mar 30. PMID 20354933
- [Background] Rademacher J, Suhling H, Greer M, Haverich A, Welte T, Warnecke G, Gottlieb J. Safety and efficacy of outpatient bronchoscopy in lung transplant recipients - a single centre analysis of 3,197 procedures. Transplant Res. 2014 May 27;3:11. doi: 10.1186/2047-1440-3-11. eCollection 2014. PMID 24917927
- [Background] Levine DJ, Glanville AR, Aboyoun C, Belperio J, Benden C, Berry GJ, Hachem R, Hayes D Jr, Neil D, Reinsmoen NL, Snyder LD, Sweet S, Tyan D, Verleden G, Westall G, Yusen RD, Zamora M, Zeevi A. Antibody-mediated rejection of the lung: A consensus report of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2016 Apr;35(4):397-406. doi: 10.1016/j.healun.2016.01.1223. Epub 2016 Feb 10. PMID 27044531
- [Background] Safavi S, Robinson DR, Soresi S, Carby M, Smith JD. De novo donor HLA-specific antibodies predict development of bronchiolitis obliterans syndrome after lung transplantation. J Heart Lung Transplant. 2014 Dec;33(12):1273-81. doi: 10.1016/j.healun.2014.07.012. Epub 2014 Jul 21. PMID 25130554
- [Background] Snyder LD, Wang Z, Chen DF, Reinsmoen NL, Finlen-Copeland CA, Davis WA, Zaas DW, Palmer SM. Implications for human leukocyte antigen antibodies after lung transplantation: a 10-year experience in 441 patients. Chest. 2013 Jul;144(1):226-233. doi: 10.1378/chest.12-0587. PMID 23328795
- [Background] Bharat A, Saini D, Steward N, Hachem R, Trulock EP, Patterson GA, Meyers BF, Mohanakumar T. Antibodies to self-antigens predispose to primary lung allograft dysfunction and chronic rejection. Ann Thorac Surg. 2010 Oct;90(4):1094-101. doi: 10.1016/j.athoracsur.2010.06.009. PMID 20868794
- [Background] Akbarpour M, Wu Q, Liu X, Sun H, Lecuona E, Tomic R, Bhorade S, Mohanakumar T, Bharat A. Clinical relevance of lung-restricted antibodies in lung transplantation. Hum Immunol. 2019 Aug;80(8):595-601. doi: 10.1016/j.humimm.2019.04.016. Epub 2019 May 8. PMID 31078336
- [Background] Emtiazjoo AM, Wilkes DS. Humoral immunity and the development of obliterative bronchiolitis after lung transplantation: is there a link? Am J Respir Cell Mol Biol. 2013 Feb;48(2):145-9. doi: 10.1165/rcmb.2012-0349RT. Epub 2012 Oct 18. PMID 23087052
- [Background] Weigt SS, Wang X, Palchevskiy V, Gregson AL, Patel N, DerHovanessian A, Shino MY, Sayah DM, Birjandi S, Lynch JP 3rd, Saggar R, Ardehali A, Ross DJ, Palmer SM, Elashoff D, Belperio JA. Gene Expression Profiling of Bronchoalveolar Lavage Cells Preceding a Clinical Diagnosis of Chronic Lung Allograft Dysfunction. PLoS One. 2017 Jan 19;12(1):e0169894. doi: 10.1371/journal.pone.0169894. eCollection 2017. PMID 28103284